CLINICAL TRIAL: NCT05308719
Title: Effect of High-Flow Nasal Therapy on Patient-Centered Outcomes in Patients at High Risk of Postoperative Pulmonary Complications After Cardiac Surgery: A Multicentre Randomised Trial
Brief Title: Nasal Oxygen Therapy After Cardiac Surgery
Acronym: NOTACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: University Hospitals, Leicester (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: P02590
Record Dates: First submitted 2021-05-08; First posted 2022-04-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Valve Disease; Coronary Artery Disease; Respiratory Failure
Keywords: High-Flow Nasal Therapy; High-Flow Nasal Oxygen; Cardiac Surgery; Pulmonary Complications
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: An adaptive, multicentre, parallel group randomised controlled clinical trial with embedded cost-effectiveness analysis.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Oxygen Therapy (No Intervention): Standard oxygen therapy arm patients will be given 30-40% inspired O2 and flow 2-6 l/min via nasal prongs or non-rebreathing mask (not humidified and not heated) post extubation. Monitoring of saturations, respiratory rate and arterial gases will happen 15 minutes post extubation and then as per local policy thereafter. If saturations < 93% then FiO2 will be increased as per respiratory escalation protocol. Standard oxygen therapy will be given for a minimum of 16 hours post extubation.
- High-Flow Nasal Therapy (Other): High-flow nasal therapy arm patients will be given AIVRO 2 high flow oxygen therapy machines post extubation, start at 30-40% inspired O2 and flow 30 l/min then up to 50 l/min over 5-10 min. Monitoring of saturations, respiratory rate and arterial gases will happen after 15 minutes post extubation and then as per local policy thereafter. If saturations < 93% then increase FiO2 as per respiratory escalation protocol. High flow nasal therapy will be given for a minimum of 16 hours post extubation.
  Interventions: Device: High Flow Nasal Therapy

INTERVENTIONS:
Device: High Flow Nasal Therapy — High Flow Nasal Oxygen (Airvo2 Device)
  Arms: High-Flow Nasal Therapy

SUMMARY:
NOTACS aims to determine if prophylactic use of high-flow nasal therapy (for a minimum of 16 hours after tracheal extubation, inclusive of up to one hour off randomised therapy for transfers around the hospital and/or physio mobilisation) increases days at home in the first 90 days after surgery, for adult patients undergoing cardiac surgery who are at high risk of postoperative pulmonary complications. The study also incorporates a health economic analysis to estimate the incremental cost-effectiveness and cost-utility of HFNT versus standard oxygen therapy at 90 days, from the view-point of the public sector, NHS and patients.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery are at significant risk of postoperative pulmonary complications that may lead to prolonged ICU and hospital stay and increase mortality. The incidence of respiratory complications may be three to four times more common in patients with intrinsic respiratory disease and lower airway obstruction (including asthma or chronic obstructive pulmonary disease (COPD)), or obese patients or current heavy smokers (> 10 pack years).

High-flow nasal therapy (HFNT) is increasingly used as a non-invasive form of respiratory support. It delivers low level, flow-dependent positive airway pressure, and is much better tolerated by patients than alternatives such as continuous positive airway pressure (CPAP) or non-invasive ventilation. Patients can talk, eat, drink and walk whilst using HFNT. However, there is equipoise regarding its prophylactic use and effect on important patient-centred outcomes. Before the intervention is recommended for routine NHS use in cardiac surgery patients at high risk of pulmonary complications, whether it improves patient-related outcomes and is cost effective in a UK setting needs to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Undergoing any elective or urgent first-time or redo cardiac surgery performed on cardiopulmonary bypass
* Have one or more clinical risk factors for postoperative pulmonary complications (COPD, asthma, lower respiratory tract infection in last 4 weeks as defined by use of antibiotics, body mass index ≥35 kg/m2 , current (within the last 6 weeks) heavy smoker (> 10 pack years)) (47, 48).

Asthma is a disease characterized by recurrent attacks of breathlessness and wheezing, and patients will have been prescribed medication by inhalers or nebulisers (either bronchodilators or steroids).

Chronic Obstructive Pulmonary Disease (COPD) is an umbrella term used to describe chronic lung diseases that cause limitations in lung airflow. The more familiar terms 'chronic bronchitis' and 'emphysema' are no longer used but are now included within the COPD 13 diagnosis. The most common symptoms of COPD are breathlessness, or a 'need for air', excessive sputum production, and a chronic cough. Patients suitable for the NOTACS study will have been prescribed medication by inhalers or nebulisers (either bronchodilators or steroids).

Exclusion Criteria:

* Requiring home oxygen therapy.
* Deep hypothermic circulatory arrest planned
* Contraindication to HFNT, e.g. nasal septal defect.
* Requirement for home ventilatory support (including: HFNT, CPAP, BiPAP)
* Requiring emergency cardiac surgery defined as surgery required within 24 hours of the decision to operate.
* Patients not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Days alive and at home without additional support in the first 90 days after surgery, for adults at high risk of postoperative pulmonary complications undergoing cardiac surgery who either receive High Flow Nasal Oxygen Therapy or Standard Oxygen Therapy | 90 days
  Number of days at home without additional support in the first 90 days after surgery (relative to baseline location and support), measured by the patient facing Patient Location and Medication Diary at 90 days
Incremental cost-effectiveness and cost-utility of High flow nasal therapy versus Standard therapy for patients undergoing cardiac surgery who are at high risk of postoperative pulmonary complications at 90 days | 90 days
  Health Economic analysis to estimate the incremental cost-effectiveness and cost-utility of High flow nasal therapy versus Standard therapy at 90 days from the view point of the public sector, NHS and patient, measured by using Patient and Family Resource Use patient facing Questionnaires at 90 days.

SECONDARY OUTCOMES:
Estimates of the incremental cost-effectiveness and cost-utility of High flow nasal therapy versus standard oxygen therapy for adult patients undergoing cardiac surgery who are at high risk of postoperative pulmonary complications at 30 days. | 30 days
  Health Economic analysis to estimate the incremental cost-effectiveness and cost-utility of High flow nasal therapy versus Standard therapy at 90 days from the view point of the public sector, NHS and patient, measured by using Patient and Family Resource Use patient facing Questionnaires at 30 days.
Incidence of mortality, pulmonary complications, intensive care re-admission rate, length of hospital and intensive care stay . | Discharge on average 7 days post operation, 30 and 90 days
  Mortality measured by the incidence of death reported from patient follow-up and medical records at 30 and 90 days.
  Incidence of postoperative pulmonary complications measured using medical notes during primary admission to hospital.
  ICU re-admission rate measured using the in-patient diary eCRF at any time during primary hospital admission Length of ICU stay (days) measured using the in-patient diary eCRF during primary hospital admission Length of hospital stay (days) measured using the in-patient diary eCRF during primary hospital admission
Incidence of major complications including sepsis, renal failure, myocardial infarction and stroke. | 30 and 90 days
  Incidence of stroke measured from patient follow-up and medical records at 30 and 90 days Incidence of sepsis measured from patient follow-up and medical records at 30 and 90 days Incidence of myocardial infarction measured from patient follow-up and medical records at 30 and 90 days
Incidence of readmission to hospital rate. | 90 days
  Incidence of readmission to hospital rate, measured using the in-patient diary eCRF during primary hospital admission and patient location and medication diary for patient completion up to 90 days
Statistical analysis of oxygenation as measured by the ROX Index (as defined as Sp02/Fi02 to respiratory rate ratio). | 2,6,12,24,and 48 hours post extubation
  Oxygenation measured by ROX Index (defined as Sp0₂/Fi0₂ to respiratory rate ratio) at 2, 6, 12, 24 and 48 hours post-extubation
Statistical analysis of patient-centered outcomes as measured using the EQ-5D-5L | Discharge on average 7 days post operation, 30 and 90 days
  Patient-reported outcomes measured using the EQ-5D-5L questionnaire at baseline, discharge, 30 and 90 days 12. Quality of Survival will be as measured using ED-5D-5L Quality adjusted life years (QALYs).
Statistical analysis of patient-centered outcomes as measured using the EQ-5D-5L Quality of Survival | Discharge on average 7 days post operation, 30 and 90 days
  Quality of Survival will be as measured using ED-5D-5L Quality adjusted life years (QALYs).
Statistical Analysis to determine if prophylactic use of high- flow nasal oxygen reduces health service and resource use. | Discharge on average 7 days post operation, 30 and 90 days
  Health service and resource use measured using Patient and Family Resource Use Questionnaires at baseline, discharge, 30 and 90 days
Statistical analysis of patient level of assistance needed with activities of daily living post surgery as measured using BARTHEL questionnaire. | Discharge on average 7 days post operation, 30 and 90 days
  Patient level of assistance needed with activities of daily living, measured using the BARTHEL questionnaire at baseline, discharge, 30 and 90 day

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Klein, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No